CLINICAL TRIAL: NCT03280238
Title: Do Pupil Dilation and Analgesia Nociception Index Reflect Pain: a Pilot Study in Healthy, Conscious Volunteers
Brief Title: Pupil Dilation and Analgesia Nociception Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Wendy Van Bogaert, Medical Student, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/278
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): * Individualized painful electrical stimuli, Surpass LT stimulator (EMS Biomedical, Korneuburg, Austria) with a bipolar felt pad electrode
  * Measurement of pupil diameter, Algiscan® (iDMed, Marseille, France)
  * Measurement of Analgesia Nociception Index, PhysioDoloris® (MetroDoloris, Lille, France)
  Interventions: Diagnostic Test: Measurement of pupil dilation and analgesia nociception index

INTERVENTIONS:
Diagnostic Test: Measurement of pupil dilation and analgesia nociception index — painful electrical stimuli of various intensities were administered to the subjects after which changes in pupil diameter and analgesia nociception index were measured

SUMMARY:
Pain assessment is crucial in clinical practice. Currently, subjective self-report is considered the most appropriate method to evaluate pain. Although several methods to assess pain objectively exist, the lack of a golden standard still remains. This pilot study assesses the changes in pupil dilation (PD) and the analgesia nociception index (ANI) as a measure of pain in healthy, conscious, male volunteers in a highly standardized and individualized environment. Nineteen subjects received three blocks of 4 individualized electrical stimulus intensities, ranging from no to severe pain. Subjects reported their perceived severity of each individual stimulus, enabling the comparison of changes in PD and ANI in relation to both administered stimulus intensities and perceived pain severities. PD and ANI were measured before and after each administration of a stimulus.

ELIGIBILITY:
Inclusion Criteria:

* good health
* no acute or chronic pain conditions
* well rested

Exclusion Criteria:

* chronic treatment
* bad health
* daily use of analgetics or other medication
* weekly tobacco use
* weekly use of recreational drugs
* more than 10 alcohol consumptions a week

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Pupil dilation in relation to pain | 2sec before until 4sec after each painful stimulus
  measurement of pupil dilation

SECONDARY OUTCOMES:
Analgesia nociception index in relation to pain | 30sec before until 60sec after each painful stimulus
  measurement of analgesia nociception index

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Van Bogaert, MS, Principal Investigator — Vrije Universiteit Brussel; Reginald Deschepper, PhD, Study Chair — Vrije Universiteit Brussel
Locations (1):
- UZ Brussel, Jette, Belgium

REFERENCES:
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Chapman CR, Oka S, Bradshaw DH, Jacobson RC, Donaldson GW. Phasic pupil dilation response to noxious stimulation in normal volunteers: relationship to brain evoked potentials and pain report. Psychophysiology. 1999 Jan;36(1):44-52. doi: 10.1017/s0048577299970373. PMID 10098379
- [Background] Koenig J, Jarczok MN, Ellis RJ, Hillecke TK, Thayer JF. Heart rate variability and experimentally induced pain in healthy adults: a systematic review. Eur J Pain. 2014 Mar;18(3):301-14. doi: 10.1002/j.1532-2149.2013.00379.x. Epub 2013 Aug 6. PMID 23922336